CLINICAL TRIAL: NCT04965402
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986166 in Healthy Japanese Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, and Drug Effects of BMS-986166 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM018-007
Record Dates: First submitted 2021-07-07; First posted 2021-07-16 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Healthy Volunteers
Keywords: BMS-986166; Japan
MeSH Terms: interventions — BMS-986166

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Panel 1: Dose 1 (Experimental)
  Interventions: Drug: BMS-986166
- Panel 2: Dose 2 (Experimental)
  Interventions: Drug: BMS-986166
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986166 — Specified dose on specified days
  Arms: Panel 1: Dose 1; Panel 2: Dose 2
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels, and drug effects of BMS-986166 in healthy Japanese male and female participants of non-childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Japanese (both biological parents are ethnically Japanese)
* Healthy as determined by medical history, physical examination, vital signs, 12-lead electrocardiograms (ECGs), and clinical laboratory evaluations
* Body Mass Index (BMI) of 18.0 to 32.0 kg/m^2, inclusive. BMI = weight (kg)/(height [m])^2

Exclusion Criteria:

* Significant acute or chronic medical illness judged to be clinically significant by the investigator and/or Sponsor's medical monitor
* History of heart disease, retinopathy, uveitis, other clinically significant ocular disease, gastrointestinal disease, stroke or transient ischemic attacks (TIA)
* Inability to tolerate oral medication
* Women who are of childbearing potential, breastfeeding, or lactating

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-02-07 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters of BMS-986166: Maximum observed blood concentration (Cmax) | Day 1, Day 28
PK parameters of BMS-986166: Time of maximum observed blood concentration (Tmax) | Day 1, Day 28
PK parameters of BMS-986166: Area under the concentration-time curve within a dosing interval (AUC(TAU)) | Day 1, Day 28
PK parameters of BMT-121795: Cmax | Day 1, Day 28
PK parameters of BMT-121795: Tmax | Day 1, Day 28
PK parameters of BMT-121795: AUC(TAU) | Day 1, Day 28

SECONDARY OUTCOMES:
Incidence of all adverse events (AEs) | Up to 77 days
Severity of all AEs | Up to 77 days
Outcome of all AEs | Up to 77 days
Incidence of all serious adverse events (SAEs) | Up to 77 days
Severity of all SAEs | Up to 77 days
Outcome of all SAEs | Up to 77 days
Severity of all AEs regardless of seriousness criteria | Up to 77 days
Investigator causality assessment of all AEs regardless of seriousness criteria | Up to 77 days
Outcomes of all AEs regardless of seriousness criteria | Up to 77 days
Incidence of clinically significant changes in physical examination findings | Up to 77 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters: PR interval | Up to 77 days
  PR interval: The time from the onset of the P wave to the start of the QRS complex
Incidence of clinically significant changes in ECG parameters: QRS interval | Up to 77 days
  QRS interval: A combination of the Q wave, R wave and S wave, the "QRS complex" represents ventricular depolarization
Incidence of clinically significant changes in ECG parameters: QT interval | Up to 77 days
  QT interval: Measured from the beginning of the QRS complex to the end of the T wave
Incidence of clinically significant changes in ECG parameters: QTcF interval | Up to 77 days
  QTcF interval: Corrected QT interval using Fridericia's formula (QTcF)
Incidence of clinically significant changes in continuous cardiac monitoring data | Up to 77 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 77 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 77 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 77 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 77 days
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 77 days
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 77 days
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 77 days
Incidence of clinically significant changes from baseline values in electrocardiogram (ECG) parameters: PR interval | Up to 77 days
Incidence of clinically significant changes from baseline values in ECG parameters: QRS interval | Up to 77 days
Incidence of clinically significant changes from baseline values in ECG parameters: QT interval | Up to 77 days
Incidence of clinically significant changes from baseline values in ECG parameters: QTcF interval | Up to 77 days
Incidence of clinically significant changes from baseline values in continuous cardiac monitoring data | Up to 77 days
Incidence of clinically significant changes from baseline values in vital signs: Body temperature | Up to 77 days
Incidence of clinically significant changes from baseline values in vital signs: Respiratory rate | Up to 77 days
Incidence of clinically significant changes from baseline values in vital signs: Blood pressure | Up to 77 days
Incidence of clinically significant changes from baseline values in vital signs: Heart rate | Up to 77 days
Incidence of clinically significant changes from baseline values in clinical laboratory results: Hematology tests | Up to 77 days
Incidence of clinically significant changes from baseline values in clinical laboratory results: Clinical Chemistry tests | Up to 77 days
Incidence of clinically significant changes from baseline values in clinical laboratory results: Urinalysis tests | Up to 77 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- West Coast Clinical Trials Global, Cypress, California, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm